CLINICAL TRIAL: NCT05000086
Title: A Pilot Study of Technetium [99Tc] Methylene Diphosphonate in the Treatment of Psoriatic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chengdu Yunke Pharmaceutical Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YK1901PsA
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Arthritis, Psoriatic
Keywords: 99Tc-MDP
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99Tc methylene diphosphonate (Experimental): 99Tc-MDP was applied as follows: for each course of treatment, 99Tc-MDP 22 mg (5.5mg/set, four sets) was injected intravenously once a day for 7 successive days, one course every 4 weeks until week 24.
  Interventions: Drug: 99Tc methylene diphosphonate

INTERVENTIONS:
Drug: 99Tc methylene diphosphonate — 22mg qd，Once a day for 7 consecutive days
  Other Names: Yunke

SUMMARY:
This study is aim to evaluate the efficacy and safety of technetium [99Tc] methylene diphosphonate (99Tc-MDP, trade name: Yunke) in the treatment of psoriatic arthritis.

DETAILED DESCRIPTION:
This is a single-arm, open label, 24 weeks study. Patients with psoriatic arthritis get 99Tc-MDP 22mg (5.5mg/set, four sets) was injected intravenously once a day for 7 successive days, one course every 4 weeks until week 24.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age;
* Clinical diagnosis of PsA according to the CASPAR classification criteria
* Active PsA at baseline defined as ≥ 3 tender joints and ≥ 3 swollen joints
* If subjects were taking csDMARDs, the doses of csDMARDs had to be stable for at least 4 weeks and had to remain the same during the trial
* The application of bDMARDs and tsDMARDs should meet the following requirements:

  1. Etanercept and its biological analogues: stop at least 4 weeks prior to their baseline visit;
  2. Other biological: stop at least 6 months prior to their baseline visit
  3. tsDMARDs: stop at least 8 weeks prior to their baseline visit
* If subjects were taking glucocorticoids, the doses of GC(prednisone < 10mg) had to be stable for at least 4 weeks and had to remain the same during the trial;
* Non steroidal anti-inflammatory drugs: if applied, the dose was stable one week prior to their baseline visit
* Negative pregnancy test for child-bearing women at screening and baseline
* Provide written informed consent

Exclusion Criteria:

* Patients with severe heart, liver, kidney and other important organ diseases
* Abnormal liver function (ALT or AST is 2 times higher than normal)
* White blood cell count less than 4,000/mm^3 (less than 4 X 10^9/L)
* Platelet count less than 100,000/mm^3 (less than 100 X 10^9/L)
* Serum creatinine more than or equal to 1.5 mg/dL (less than or equal to 132.6 μmol/L)
* Pregnancy or breastfeeding women
* Contraindications to 99Tc-MDP therapy and/or known hypersensitivity to 99Tc-MDP
* Participated in other drugs clinical trials within 4 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients Achieving DAS28-CRP<=3.2 | 24 weeks
  DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. DAS28-CRP score of <=3.2 indicates low disease activity. <2.6 means disease remission
Proportion of Patients Achieving DAS28-ESR<=3.2 | 24 weeks
  DAS28-ESR: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (ESR) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. DAS28-ESR score of <=3.2 indicates low disease activity. <2.6 means disease remission

SECONDARY OUTCOMES:
Change in PASI From Baseline From Baseline | 24 weeks
  Psoriasis Area and Severity Index
Change in HAQ-DI Score From Baseline | 24 weeks
  The HAQ-DI is a standardized measure of physical function in arthritis. The HAQ-DI questionnaire contains 20 items divided into 8 domains that measure: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability.
ACR20 | 12 weeks
  The ACR is a standard criteria originally developed to measure the effectiveness of various arthritis medications or treatments in clinical trials for RA, but is also widely used in PsA. The ACR measures improvement in tender joint count (TJC) or swollen joint count (SJC), and improvement in at least 3 of the following 5 parameters: Patient Global Assessment (PtGA), Physician's Global Assessment of Disease Activity (PhGA), physical function (using HAQ-DI) and acute phase reactant (using CRP). ACR 20 response is achieved if ≥ 20% improvement in tender joint count (TJC) or swollen joint count (SJC) as well as a ≥ 20%/≥ 50%/≥ 70% improvement in ≥ 3 of the other 5 parameters.
Change in Disease Activity in Psoriatic Arthritis Score (DAPSA) Score From Baseline | 24 weeks
  Disease Activity in Psoriatic Arthritis Score (DAPSA) score is a the sum of swollen joint count (66 joints), tender joint count (68 joints), CRP (mg/dL), Patient's Assessment of Pain (on a 10-unit VAS;0=no pain, 10=worst possible pain), and Patient's Global Assessment of Disease Activity (arthritis, on a 10-unit VAS; 0 to 100 centimeter [cm] VAS, 0=excellent and 10=poor). Change from baseline in DAPSA measures the change in disease activity, where a negative change indicates an improvement and a positive change indicates worsening of disease activity.
Percentage of Participants in MDA | 24 weeks
  MDA for PsA was defined as fulfilling at least 5 of the following 7 criteria: TJC ≤ 1 (out of TJC68 assessed in this study), SJC ≤ 1 (out of SJC66 assessed in this study), PASI ≤ 1 or BSA ≤ 3; Patient's assessment of pain VAS ≤ 15, PtGA VAS ≤ 20, HAQ-DI score ≤ 0.5, and tender entheseal points ≤ 1
Change in Tender Joint Count (TJC) 68 from baseline | 12 weeks and 24 weeks
  TJC is determined by physical examination of 68 joint counts that are assessed for tenderness.
Change in Swollen Joint Count (SJC) 66 from baseline | 12 weeks and 24 weeks
  SJC is determined by physical examination of 66 joint counts that are classified as either swollen or not swollen.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College hospital, Beijing, Dongcheng, China

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years after article publication
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to lpumch@126.com. To gain access, data requestors will need to sign a data access agreement

REFERENCES:
- [Background] Shen S, Wang W, Yang C, Xu B, Zeng L, Qian Y. Effect of technetium-99 conjugated with methylene diphosphonate (99 Tc-MDP) on OPG/RANKL/RANK system in vitro. J Oral Pathol Med. 2019 Feb;48(2):129-135. doi: 10.1111/jop.12801. Epub 2018 Dec 9. PMID 30421571
- [Background] Mu R, Liang J, Sun L, Zhang Z, Liu X, Huang C, Zhu P, Zuo X, Gu J, Li X, Li X, Liu Y, Feng P, Li Z. A randomized multicenter clinical trial of 99 Tc-methylene diphosphonate in treatment of rheumatoid arthritis. Int J Rheum Dis. 2018 Jan;21(1):161-169. doi: 10.1111/1756-185X.12934. Epub 2017 Feb 3. PMID 29356462
- [Background] Fu Q, Feng P, Sun LY, Zuo XX, Zhao DB, He DY, Wu HX, Zhang W, Zhang W, Du F, Bao CD. A double-blind, double-dummy, randomized controlled, multicenter trial of 99Tc-methylene diphosphonate in patients with moderate to severe rheumatoid arthritis. Chin Med J (Engl). 2021 May 19;134(12):1457-1464. doi: 10.1097/CM9.0000000000001527. PMID 34039871
- [Background] Su D, Shen M, Gu B, Wang X, Wang D, Li X, Sun L. (99) Tc-methylene diphosphonate improves rheumatoid arthritis disease activity by increasing the frequency of peripheral gammadelta T cells and CD4(+) CD25(+) Foxp3(+) Tregs. Int J Rheum Dis. 2016 Jun;19(6):586-93. doi: 10.1111/1756-185X.12292. Epub 2014 Jan 28. PMID 24467668